CLINICAL TRIAL: NCT04189406
Title: Turner Syndrome Minipuberty Study A Prospective, Descriptive Cohortstudy
Brief Title: Turner Syndrome Minipuberty Study
Acronym: Minipuberty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-5955
Record Dates: First submitted 2019-11-25; First posted 2019-12-06 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-03

CONDITIONS: Turner Syndrome; Infertility, Female; Premature Ovarian Failure; Gonadal Dysgenesis; Premature Menopause; Sex Chromosome Disorders; Ovarian Diseases
Keywords: Minipuberty; Turner Syndrome; Infertility; Premature Ovarian Failure
MeSH Terms: conditions — Turner Syndrome; Infertility, Female; Primary Ovarian Insufficiency; Gonadal Dysgenesis; Menopause, Premature; Sex Chromosome Disorders; Ovarian Diseases; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Analysing LH, FSH, AMH, estradiol, inhibin B and testosterone in plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Girls with Turner syndrome: Girls with a pre- or perinatal diagnosis TS who are born in a medical centre in the Netherlands during the duration of the study.
  The subjects will have an extra venapuncture of 3.5 mL blood at 3 and 9 months.
  Interventions: Other: Venapunction

INTERVENTIONS:
Other: Venapunction — A blood sample of 3.5 mL (0.2 mL serum for FSH and LH, 0.15 mL serum for E2, 0.15 mL serum for T, 0.15 mL serum for AMH and 0.25 mL serum for Inhibin B) will be collected of all girls with TS at 3 months and 9 months of age. For the girls with TS, this will be collected with an extra venapuncture during a regular outpatient visit within the usual care.

SUMMARY:
Rationale: Due to accelerated germ cell loss, infertility is a major problem in girls with Turner syndrome (TS). Therefore, cryopreservation of ovarian tissue or oocytes before exhaustion of the ovarian reserve may preserve fertility in patients with TS. However, in the majority of females with TS , the ovarian reserve is exhausted before the age of menarche. Early markers indicating and predicting the ovarian reserve are necessary. During mid-childhood the hypothalamic-pituitary-gonadal (HPG) axis is quiescent and gonadotropins are usually unmeasurable. Nonetheless, this axis is active during infancy. Therefore, gonadotropins are measurable with peak values at 3 months of age and with lower (but still measurable) values at 9 months of age, in a period called the minipuberty. The aim of this study is to find markers of ovarian capacity, during the minipuberty, in order to predict ovarian reserve in the future.

Objective: The hormonal range of LH, FSH, AMH, inhibin B, testosterone and estradiol in girls with TS during the minipuberty and the relation of the hormone serum levels with the karyotype.

Study design: A prospective, cohort study with a duration of 3 years. Study population: Girls with a pre- or perinatal diagnosis TS who are born in a medical centre in the Netherlands during the duration of the study

Main study parameters/endpoints: Serum levels of FSH, LH, AMH, inhibin B, testosterone and estradiol at the age of 3 and 9 months.

DETAILED DESCRIPTION:
Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The subjects will have twice an extra venapunction for collection of 3.5mL blood during their infancy, which is not stated in the guidelines for TS. There is very little risk for adverse events associated with this blood sample collection, however it is an extra procedure. The outcome parameters will not be helpful for individual study participants, however they are likely to help clinicians and researchers in understanding how the ovarian function operates develops in girls with TS. Furthermore, these markers could be used to estimate the ovarian reserve and the urgency of fertility preservation in young females with TS. This information could help clinicians, patients and their parents in decision making.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in the TS group of this study, a subject must meet all of the following criteria:

* A diagnosis of TS before the age of three months;
* Girls with a diagnosis of classic TS or other variants (i.e. 45,X, 45,X/46XiXq, 45,X/46,XY, 45,X/46,XX, 45,X/47,XXX, 45,X/46,X,r(X), 46,XiXq, other);
* Whose parents have agreed to participate in the study through a signed written informed consent form.

In order to be eligible to participate in the control group of this study, a subject must meet all of the following criteria:

* No diagnosis of TS or any other diagnosis that might affect the HPG axis;
* Girls that will have a blood collection within their usual care at 3 months and at 9 months of age.
* Whose parents have agreed to participate in the study through a signed informed consent form.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Any other diagnosis besides TS that might affect the HPG axis;
* Ovarian surgery in the medical history;
* Critical illness;
* The use of medication affecting the HPG axis (e.g. estrogen suppletion therapy)

Ages: 1 Month to 3 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We include girls with the diagnosis TS before the age of 3 months based on full or partial absence of one X-chromosome or a mosaic pattern. We will recruit the girls with TS from all medical centres in the Netherlands. The control group consists of girls who have blood collected at 3 months and at 9 months of age for another indication. Participants in the control group will be recruited in the Radboudumc in Nijmegen.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Defining the LH range in blood during minipuberty in girls with TS at 3 months of age and at 9 months of age | 1 year after venapuncture
  LH (luteinizing hormone) will be collected with a venapuncture and analysed with the Elecsys method on the Cobas E801system of Roche.
Defining the FSH range during minipuberty in girls with TS at 3 months of age and at 9 months of age | 1 year after venapuncture
  FSH (follicle stimulating hormone) will be collected with a venapuncture and analysed with the Elecsys method on the Cobas E801system of Roche.
Defining the AMH range during minipuberty in girls with TS at 3 months of age and at 9 months of age | 1 year after venapuncture
  AMH (Anti-Müllerian hormone) will be collected with a venapuncture and analysed on the Access of Beckman Coulter.
Defining the estradiol range during minipuberty in girls with TS at 3 months of age and at 9 months of age | 1 year after venapuncture
  estradiol will be collected with a venapuncture and analysed with the LCMSMS analysis method.
Defining the testosterone range during minipuberty in girls with TS at 3 months of age and at 9 months of age | 1 year
  testosterone will be collected with a venapuncture and analysed with the LCMSMS analysis method.
Defining the inhibin B range during minipuberty in girls with TS at 3 months of age and at 9 months of age | 1 year after venapuncture
  inhibin B will be collected with a venapuncture and analysed with the GEN II ELISEA of Beckman Coulter.

SECONDARY OUTCOMES:
Patient's karyotype vs LH | 1 year after venapuncture
  The association between patient's karyotype and LH level at 3 months of age and 9 months of age
Patient's karyotype vs FSH | 1 year after venapuncture
  The association between patient's karyotype and FSH level at 3 months of age and 9 months of age
Patient's karyotype vs AMH | 1 year after venapuncture
  The association between patient's karyotype and AMH level at 3 months of age and 9 months of age
Patient's karyotype vs estradiol | 1 year after venapuncture
  The association between patient's karyotype and estradiol level at 3 months of age and 9 months of age
Patient's karyotype vs testosterone | 1 year after venapuncture
  The association between patient's karyotype and testosterone level at 3 months of age and 9 months of age
Patient's karyotype vs inhibin B | 1 year after venapuncture
  The association between patient's karyotype and inhibin B level at 3 months of age and 9 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Janielle vd Velden, MD, PhD, Principal Investigator — Paediatric endocrinologist, Radboudumc, Nijmegen
Locations (13):
- Righospitalet, University of Copenhagen, Copenhagen, Denmark
- Germany (3):
  - Universitätsklinikum der Ruhr-Universität Bochum, Bochum
  - Justus-Liebig Universität Giessen, Giessen
  - Universitätsklinikum Tübingen, Tübingen
- Netherlands (7):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Amsterdam University medical center, Amsterdam
  - University medical center Groningen, Groningen
  - Leiden University medical center, Leiden
  - Maastricht University medical center, Maastricht
  - Erasmus University medical center, Rotterdam
  - University medical Center Utrecht, Utrecht
- Medical university of Silesia, Katowice, Poland
- University hospital of Umea, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernard V, Donadille B, Zenaty D, Courtillot C, Salenave S, Brac de la Perriere A, Albarel F, Fevre A, Kerlan V, Brue T, Delemer B, Borson-Chazot F, Carel JC, Chanson P, Leger J, Touraine P, Christin-Maitre S; CMERC Center for Rare Disease. Spontaneous fertility and pregnancy outcomes amongst 480 women with Turner syndrome. Hum Reprod. 2016 Apr;31(4):782-8. doi: 10.1093/humrep/dew012. Epub 2016 Feb 13. PMID 26874361
- [Background] Borgstrom B, Hreinsson J, Rasmussen C, Sheikhi M, Fried G, Keros V, Fridstrom M, Hovatta O. Fertility preservation in girls with turner syndrome: prognostic signs of the presence of ovarian follicles. J Clin Endocrinol Metab. 2009 Jan;94(1):74-80. doi: 10.1210/jc.2008-0708. Epub 2008 Oct 28. PMID 18957497
- [Background] Bryman I, Sylven L, Berntorp K, Innala E, Bergstrom I, Hanson C, Oxholm M, Landin-Wilhelmsen K. Pregnancy rate and outcome in Swedish women with Turner syndrome. Fertil Steril. 2011 Jun 30;95(8):2507-10. doi: 10.1016/j.fertnstert.2010.12.039. Epub 2011 Jan 22. PMID 21256486
- [Background] Burgoyne PS, Baker TG. Perinatal oocyte loss in XO mice and its implications for the aetiology of gonadal dysgenesis in XO women. J Reprod Fertil. 1985 Nov;75(2):633-45. doi: 10.1530/jrf.0.0750633. PMID 3906118
- [Background] Fechner PY, Davenport ML, Qualy RL, Ross JL, Gunther DF, Eugster EA, Huseman C, Zagar AJ, Quigley CA; Toddler Turner Study Group. Differences in follicle-stimulating hormone secretion between 45,X monosomy Turner syndrome and 45,X/46,XX mosaicism are evident at an early age. J Clin Endocrinol Metab. 2006 Dec;91(12):4896-902. doi: 10.1210/jc.2006-1157. Epub 2006 Sep 12. PMID 16968797
- [Background] Huang JY, Tulandi T, Holzer H, Lau NM, Macdonald S, Tan SL, Chian RC. Cryopreservation of ovarian tissue and in vitro matured oocytes in a female with mosaic Turner syndrome: Case Report. Hum Reprod. 2008 Feb;23(2):336-9. doi: 10.1093/humrep/dem307. Epub 2007 Dec 2. PMID 18056118
- [Background] Johannsen TH, Main KM, Ljubicic ML, Jensen TK, Andersen HR, Andersen MS, Petersen JH, Andersson AM, Juul A. Sex Differences in Reproductive Hormones During Mini-Puberty in Infants With Normal and Disordered Sex Development. J Clin Endocrinol Metab. 2018 Aug 1;103(8):3028-3037. doi: 10.1210/jc.2018-00482. PMID 29917083
- [Background] Lanciotti L, Cofini M, Leonardi A, Penta L, Esposito S. Up-To-Date Review About Minipuberty and Overview on Hypothalamic-Pituitary-Gonadal Axis Activation in Fetal and Neonatal Life. Front Endocrinol (Lausanne). 2018 Jul 23;9:410. doi: 10.3389/fendo.2018.00410. eCollection 2018. PMID 30093882
- [Background] Pasquino AM, Passeri F, Pucarelli I, Segni M, Municchi G. Spontaneous pubertal development in Turner's syndrome. Italian Study Group for Turner's Syndrome. J Clin Endocrinol Metab. 1997 Jun;82(6):1810-3. doi: 10.1210/jcem.82.6.3970. PMID 9177387
- [Background] Stochholm K, Juul S, Juel K, Naeraa RW, Gravholt CH. Prevalence, incidence, diagnostic delay, and mortality in Turner syndrome. J Clin Endocrinol Metab. 2006 Oct;91(10):3897-902. doi: 10.1210/jc.2006-0558. Epub 2006 Jul 18. PMID 16849410
- [Background] Sutton EJ, McInerney-Leo A, Bondy CA, Gollust SE, King D, Biesecker B. Turner syndrome: four challenges across the lifespan. Am J Med Genet A. 2005 Dec 1;139A(2):57-66. doi: 10.1002/ajmg.a.30911. PMID 16252273